CLINICAL TRIAL: NCT01518881
Title: A Placebo-Controlled, Single-Blind, Single-Ascending Dose Study With Additional Multiple-Ascending Dose Cohorts to Evaluate the Safety, Tolerability and Pharmacokinetics of TKM-100201 in Healthy Human Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetic First in Human (FIH) Study of Intravenous (IV) TKM-100201 Infusion
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Corporate decision to reformulate the investigational product.
Sponsor: Arbutus Biopharma Corporation (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TKM-EBOV-001
Record Dates: First submitted 2011-11-08; First posted 2012-01-26 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Ebola Virus Infection
MeSH Terms: conditions — Hemorrhagic Fever, Ebola | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TKM-100201 (Experimental)
  Interventions: Drug: TKM-100201
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TKM-100201 — IV Infusion
  Other Names: TKM-Ebola
  Arms: TKM-100201
Drug: Placebo — IV infusion
  Other Names: Normal Saline
  Arms: Placebo

SUMMARY:
This is a phase 1, single-center, placebo-controlled, single-blind, first-in-human, single-ascending dose study with additional multiple-ascending dose cohorts in healthy male and female volunteers.

DETAILED DESCRIPTION:
A maximum of 56 healthy adult (male and female) subjects will participate in this study, in two stages. In Stage 1, the Single-Ascending Dose (SAD) phase of the study will have up to six cohorts with 4 subjects (3 receiving TKM-100201 and 1 receiving saline placebo) in each cohort. Additional cohorts may be enrolled if a maximum tolerated dose (MTD) is not established after the initial six cohorts. In Stage 2, the Multiple-Ascending Dose (MAD) portion of the study will have up to three cohorts with four subjects (3 receiving TKM-100201 and 1 receiving saline placebo) in each cohort. Additional cohorts may be enrolled if a maximum tolerated dose (MTD) is not established after the initial three cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Informed of the nature of the study and have agreed to and are able to read, review and sign the informed consent document at screening. The informed consent document will be written in English, therefore the volunteer must have the ability to read and communicate in English.
2. Able to comply with all protocol-specified visit schedules and requirements.
3. Completed the screening process within 14 days prior to dosing.
4. Healthy male and female volunteers 18 to 50 years of age, inclusive, at the time of dosing.
5. Body mass index (BMI) between 22 kg/m2 to 35 kg/m2, inclusive, and weigh at least 110 lbs.
6. Judged by an Investigator to be in good health as documented by the medical history, physical examination (including but may not be limited to an evaluation of the cardiovascular, gastrointestinal, respiratory and central nervous systems), vital sign assessments, 12-lead ECG, clinical laboratory assessments, and by general observations. Any abnormalities or deviations outside the normal ranges for any of clinical testing (laboratory tests, ECG, vital signs) can be repeated at the discretion of the Investigator(s) and judged to be not clinically significant for study participation.
7. Adequate hepatic, renal, hematologic and clotting function as defined by total bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), serum creatinine, D-dimer and International normalized ratio (INR) within normal range as determined by the Investigator(s) and Sponsor Medical Monitor.
8. Female volunteers must be one of the following:

   * naturally postmenopausal (no menses) for > 2 years and has a documented FSH level >40 mIU/mL; or
   * have a documented history of ovarian failure; or
   * surgically postmenopausal (bilateral oophorectomy or hysterectomy). Female volunteers that are surgically postmenopausal must provide documentation of the bilateral oophorectomy or hysterectomy prior to Day 1 dosing to be eligible for participation in the study; or
   * Women of childbearing potential (FSH ≤40 mIU/mL) must have negative serum hCG at screening, a negative urine pregnancy test prior to the first study treatment, and must agree to utilize highly effective contraception methods (two separate forms of contraception, one of which must be an effective barrier method, or be non-heterosexually active, or have a vasectomized partner) from screening throughout the duration of study treatment and for 1 month after the last administration of investigational product.
9. Male volunteers who are sexually active must be willing to use effective barrier contraception (e.g., condom with spermicide) during heterosexual intercourse from screening throughout the duration of study treatment and for 1 month after the last dose of investigational product.

Exclusion Criteria:

1. Evidence or history of clinically significant hematologic, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic or allergic disease at screening or medication for comorbidity which, in dialogue between the Investigator and Medical Monitor would preclude subject participation in the clinical trial.
2. Reports an uncontrolled psychiatric disorder or neurologic disease or seizure disorder not controlled by medication.
3. Subject has a history of existing clinically significant cardiovascular disease (for example, uncontrolled hypertension, unstable angina, congestive heart failure or serious cardiac arrhythmias). In addition New York Heart Association Functional Classification Class II or greater will be excluded (see Appendix).
4. Reports history of coronary heart disease (CHD), CHD-equivalent disease or CHD risk >20% as designated by the National Cholesterol Education Program Adult Treatment Panel III.
5. Current diagnosis or known history of liver disease (e.g. acute or chronic hepatitis or liver cirrhosis).
6. Presence of any clinically significant results from laboratory tests, vital signs assessments and ECGs as judged by the Investigator(s).
7. Reports receiving any antiviral drugs, investigational drugs, biologics, or devices within 28 days prior to study treatment or planned use during the course of the study.
8. Reports receiving naturopathic medications, herbal supplements, or lipid lowering therapies within 28 days prior to study treatment of planned use during the course of the study.
9. Recent treatment with alternative therapies which, in the view of the Investigator(s) or the Medical Monitor, could potentially confound clinical and laboratory assessments.
10. Demonstrates a marked baseline prolongation of QT/QTc interval (e.g. repeated demonstration of a QTc interval >450 ms)
11. Reports concomitant use of any medication that prolongs the QT/QTc interval.
12. Reports a history of additional risk factors for torsades de pointes (e.g. heart failure, hypokalemia, family history of Long QT Syndrome).
13. When confirmed upon additional testing, demonstrates a reactive screen for hepatitis B surface antigen, hepatitis C antibody, or HIV antibody.
14. Reports infections requiring antibiotic therapy within 30 days of screening (as determined by the Investigator[s]).
15. Reports a history of Ebola virus exposure.
16. Reports an occupational health risk of exposure to Ebola virus known to be higher than that of the general population.
17. Reports a known or suspected hypersensitivity or previous severe reactions to any of the constituents of the investigational product including oligonucleotide- or lipid-based products, liposomal drug products, and phospholipid-based products (parenteral nutrition, Intralipid).
18. Reports a history of clinically significant allergies including food or drug allergies.
19. Demonstrates a positive drug or alcohol screen.
20. Reports a history of drug or alcohol addiction or abuse within the past 1 year.
21. Subject is unwilling to limit alcohol consumption during the study (males: 2 drinks/day [30 g], <12 drinks/week [120 g] and females: 2 drinks/day [20 g], <12drinks/week [120 g]).
22. Reports donating blood within 28 days prior to dosing. All volunteers will be advised not to donate blood for four weeks after completing the study.
23. ports donating plasma (eg, plasmapheresis) within 14 days prior to dosing. All volunteers will be advised not to donate plasma for four weeks after completing the study.
24. Demonstrates, in the opinion of study staff, veins unsuitable for repeated venipuncture or IV infusion (eg, veins difficult to locate, access, or puncture; veins with a tendency to rupture during or after puncture).
25. Reports being capable of becoming pregnant, breastfeeding, or lactating.
26. Demonstrates a positive pregnancy screen.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of Treatment with TKM-100201 | 1 month
  Subjects will be monitored for treatment-emergent and dose-limiting toxicity (DLT). If there are any adverse events (changes from baseline in laboratory parameters, vitals and/or infusion reactions) during these monitoring periods, the Independent Safety Committee, will discuss the dosing of the remaining subjects.
  Before proceeding to the next dose cohort, the Independent Safety Committee will evaluate whether dose escalation will be permitted based on demonstration of adequate safety and tolerability.

SECONDARY OUTCOMES:
Pharmacokinetics - Cmax, Tmax and AUC will be calculated | 29 days post infusion
  Time-points: Before infusion, mid-point of infusion, end of infusion and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48 hours after infusion and day 7, day 10, day 15, day 22 and day 29.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory M Haugen, M.D., Principal Investigator — Cetero Research, San Antonio
Locations (1):
- Cetero Research, Fargo, North Dakota, United States